CLINICAL TRIAL: NCT07025200
Title: Effect of Dupilumab on Mucus Plugs and Inflammatory Patterns in Severe Asthmatic Patients - a Pilot Study
Brief Title: DETACT sEvere asThmAtiC paTients - a Pilot Study
Acronym: DETACT
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Marco Idzko, Univ. Prof. Dr., Medical University of Vienna
Other Study IDs: 1741/2022
Record Dates: First submitted 2024-02-02; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — dupilumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — For the purpose of the study we will collect blood samples as well as bronchoscopy-derived samples as bronchoalveolar lavage (BAL) fluid, bronchial lining fluid and bronchial biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Dupilumab treated patients: All patients will be administered subcutaneous doses of dupilumab every 2 weeks.
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — Clinical assessment, lung function, CT-scans and Bronchoscopy prior to and 22 weeks after initiation of Dupilumab.

SUMMARY:
The objective of this study is to investigate the effect of dupilumab treatment on mucus plugging in severe asthma patients with severe eosinophilic asthma. Therefore, the investigators plan to apply computer tomography to investigate mucus plugging and thoroughly examine different airway samples from Type 2-high severe asthmatic patients at a cellular, molecular, microbiological and metabolomic level. This study will help to unravel underlying treatment mechanisms of dupilumab therapy in severe asthmatics.

DETAILED DESCRIPTION:
In this prospective exploratory pilot study, the objective is to enroll 10 participants with severe asthma who are candidates for Dupilumab treatment. The study's individual duration will not exceed 26 weeks. Before enrollment, informed consent will be obtained from all subjects. All patients with severe Type 2 Asthma can be included according to inclusion- and exclusion criteria. Those with a history of monoclonal antibody treatment for asthma may be included after a washout period of 2 half-lives or 1 month (whichever is longer).

Prior to commencing Dupilumab, the investigators will assess patient-reported outcomes using the Asthma Control Questionnaire (ACQ-6), Asthma Control Test (ACT), and mini Asthma Quality of Life Questionnaire (miniAQLQ). Additionally, the investigators will review concomitant medication, conduct Spirometry, measure fraction of exhaled nitric oxide (FeNO), perform ultra high-resolution computer tomography of the lungs, draw blood for laboratory samples, and carry out bronchoscopy with bronchoalveolar lavage and biopsies.

Subsequently, Dupilumab treatment will be initiated, and patients will visit our center every 2 weeks for clinical assessments, including monitoring adverse events, lung function, laboratory samples, and Dupilumab administration. After 22 weeks, the investigators will repeat computer tomography of the lungs and bronchoscopy. For patients who do not experience clinical improvement, Dupilumab treatment will be discontinued after 6 months.

ELIGIBILITY:
Inclusion Criteria:

All patients who:

* are ≥18 years of age
* have a recorded clinical diagnosis of asthma (ICD-10 Code: J45)
* meet the requirements for treatment of severe T2-high asthma for Dupilumab defined as:
* FeNO > 25 ppB
* two measurements of at least 250 eosinophils /µl in the blood OR one measurement of blood eosinophils at least 250 cells/µl during reduction of OCS dosing if treated with oral corticosteroids and/or one measurement of sputum ≥ 2% or BAL eosinophils ≥ 1%
* have a history of treatment with monoclonal antibodies for asthma if a wash out period of 2 half-lives or 1 month (whatever is longer) has passed

Exclusion Criteria:

Patients who:

* are pregnant as determined by a ß-HCG test
* have severe anatomic variations or deviations that do not allow bronchoscopy
* suffer from additional others confounding underlying lung disorder including but not limited to: Bronchiectasis, chronic obstructive pulmonary disorder (COPD), pulmonary fibrosis, emphysema, Cystic fibrosis, any known parasitic infections and lung cancer.
* show pulmonary conditions with symptoms of asthma and blood eosinophilia, including but not limited to: Churg-Strauss syndrome, allergic bronchopulmonary aspergillosis, hypereosinophilic syndrome
* suffer from a mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study,
* have clinically meaningful comorbidity as determined by the evaluating committee,
* experience of an asthma exacerbation within 4 weeks prior to the first main visit
* immune disorder and/or immunosuppressive treatment (e.g. cyclosporine), ongoing biological treatment of asthma (e.g., mepolizumab, omalizumab, benralizumab) or last biological treatment 2 half-lives or 1 month before the first main visit
* have a history of drug and alcohol abuses
* are currently smoking or are former smokers for less than 6 months with >10 pack years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe Type 2 asthma for whom Dupilumab therapy is indicated.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Effect of Dupilumab treatment on mucus plugging in patients with severe eosinophilic asthma | 26 weeks
  CT scans of the lungs will be done on baseline and 22 weeks after begin applying ultra-high resolution CT technique (special resolution 0.2 mm). The examinations will be performed as no-contrast CTs in sustained deep inspiration and expiration. The images will be investigated and scored independently by two thoracic radiologists. Both radiologists will score the extent of air-trapping, bronchial wall thickening and mucus plugging per pulmonary segment based on the following scale:
  * absent (0)
  * minimal (1)
  * moderate (2)
  * extensive (3) Prior to the evaluation of study scans, both radiologists will undergo a consensus reading on CT scans not included in the study.

SECONDARY OUTCOMES:
Change in asthma control | 26 weeks
  We will assess change in asthma control under Dupilumab treatment using the Asthma Control Test (ACT), Asthma Control Questionnaire-6 (ACQ-6) and mini Asthma Quality of Life Questionnaire (mAQLQ).
Change in number of asthma exacerbations | 26 weeks
  Asthma exacerbations will be defined as events requiring the use of systemic corticosteroids for at least three consecutive days.
Change in peripheral blood eosinophil count (PBEC) | 26 weeks
  PBEC, measured in cells per microliter (cells/µL), will be assessed every two weeks at the clinic.
Change in forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC) | 26 weeks
  FEV₁ and FVC, expressed in milliliters (mL) and as percentages of the predicted values, will be assessed during clinic visits. Additionally, patients will receive home spirometry devices to enable more frequent lung function monitoring between appointments
Change in fractional exhaled nitric oxide (FeNO) | 26 weeks
  FeNO will be measured daily at home using portable devices, as well as every two weeks at the clinic. Measurements will be expressed in parts per billion (ppb).
Change in Cellular Composition and Activation | 26 weeks
  Characterization of immune cell populations and their activation states isolated from bronchoalveolar lavage (BAL) cells.
Change in Inflammatory Mediators | 26 weeks
  Quantification of inflammatory mediator concentrations in BAL supernata
Change in Transcriptional Profiling | 26 weeks
  Analysis of gene expression profiles in BAL cells and lung tissue using transcriptional sequencing techniques.
Lung Microbiome | 26 weeks
  Assessment of microbial community composition in BAL samples.
Metabolomic Profile | 26 weeks
  Characterization of metabolite composition in BAL fluid.

OTHER OUTCOMES:
Safety and Tolerability | 26 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Clinic of Internal Medicine II, Department of Pulmonology, Vienna, Vienna, Austria